CLINICAL TRIAL: NCT04170270
Title: Oral Versus Intravenous Omeprazole in Management of Bleeding Peptic Ulcer: Randomized Controlled Trial
Brief Title: Oral Omeprazole in Bleeding Peptic Ulcer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Zeinab Nasr El Din Ahmed, Principle Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: bleeding peptic ulcer
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Bleeding Peptic Ulcer
MeSH Terms: conditions — Peptic Ulcer Hemorrhage | interventions — Omeprazole

STUDY DESIGN:
Intervention Model Description: comparison between oral and intravenous omeprazole in management of bleeding peptic ulcer
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oral omeprazole (Experimental): oral omeprazole in bleeding peptic ulcer after endoscopic therapy 40 mg twice daily for 72 hours
  Interventions: Drug: Omeprazole
- intravenous omeprazole (Active Comparator): intravenous omeprazole in bleeding peptic ulcer after endoscopic therapy as continuous infusion at rate of 8 mg/hour for 72 hours
  Interventions: Drug: Omeprazole

INTERVENTIONS:
Drug: Omeprazole — Pre endoscopically: all patients will receive 80 mg omeprazole by 30 minute IV infusion.
  After performing upper endoscopy (with initial hemostasis), the patient will be randomly allocated into two groups; group A patients will receive oral omeprazole, while group B patients are intended to receive IV omeprazole.
  For patients of group A, omeprazole 40 mg will be administrated orally every 12 hours for 72 hours. Regarding group B, continuous infusion of omeprazole will be administrated at a rate of 8 mg/hour, for 72 hours.

SUMMARY:
Find out if there is a significant difference between clinical outcome among the patients with bleeding peptic ulcer treated with oral omeprazole compared to those treated with intravenous omeprazole.

DETAILED DESCRIPTION:
Globally, Peptic ulcer disease is the most common cause of upper gastrointestinal bleeding (UGIB), accounting for about 50% of cases. It remains a serious medical problem with significant morbidity and mortality (1, 2). However, in Egypt, bleeding peptic ulcer comes second to the bleeding varices in order of frequency (approximately 30%) (3).

Over the past 20 years, mortality resulting from bleeding peptic ulcer significantly decreased through researches on primary endoscopic hemostasis, due to improvement in pre- and post-endoscopic management, as well as identification of patients at a risk of catastrophic events-for close observation and focused intensive management (4).However, the risk of patients with bleeding peptic ulcers significantly increased owing to the aging population with multiple comorbidities, as well as the increasing use of aspirin and non-steroidal anti-inflammatory drugs (5).

Endoscopic therapy significantly reduces further bleeding, surgery, and mortality in patients with bleeding peptic ulcer and is now recommended as the first hemostatic modality for these patients. However, there is a high risk of peptic ulcer re-bleeding in 14-36% of patients, in spite of efficient endoscopic intervention (6).

Intravenous proton pump inhibitors (PPIs) are effective as adjuvant pharmacotherapy in preventing re-bleeding in these patients (7).

Gastric acid inhibits clot formation and promotes clot lyses and accordingly, disturbs hemostasis of ulcers in the stomach and duodenum (8). Therefore, reduction of gastric acid secretion can prevent ulcer re-bleeding.

The use of high-dose intravenous PPIs is standard practice in the management of upper gastrointestinal bleeding (9).

High dose IV PPI has faster adequate acid suppression effect (gastric acid PH > 6) than high dose oral PPI . In addition, Compared to standard dose of oral PPI, high dose oral PPI has faster acid suppression (10, 11). However, the optimal route, dose, and duration of PPI therapy after endoscopic therapy of a bleeding peptic ulcer remain controversial.

UGIB continues to represent a signiﬁcant clinical and economic burden to society. Intravenous PPI therapy is more expensive than oral one. Therefore, the therapy has to be assessed from a cost-effectiveness perspective (12).

Several controlled trials and meta-analyses have shown the comparable efficacy of IV and oral PPI in treating ulcers at high risk of re-bleeding after endoscopic therapy. However, further studies to confirm their results were recommended (13, 14).

The investigators will evaluate and compare the efficacy and safety profile of oral PPI compared to IV PPI in preventing re-bleeding from peptic ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Peptic ulcer of the esophagus (lower part), stomach, and duodenum with one or more endoscopic signs of high risk for re-bleeding (ulcer bed exhibiting active bleeding (spurting/oozing), non-bleeding visible vessel, and adherent clot).

Exclusion Criteria:

* Pregnant patients.
* Pediatric patients (less than 18 years).
* Ulcer with endoscopic signs suspicious of neoplastic disease (greater than 3 cm, irregular shape, uneven base, irregular edges, moth eaten appearance of peri ulcer folds, associated with a mass)
* Use of PPI 14 days or less before enrollment.
* Other sources of UGIB.
* Bleeding tendency (platelet count <50,000/mL, prothrombin time > 14 sec, prothrombin concentration <30%, anticoagulant therapy)
* Uremia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
recurrent bleeding | 15 days
  Re-bleeding will be suspected if hematemesis or melena recur or of the patient develop one or more of the following: orthostatic hypotension, unstable vital signs (systolic blood pressure< 90 mmHg and pulse rate> 120/min), reduction of hemoglobin level> 2 gm/dL (despite blood transfusion), during 24 hour period.

SECONDARY OUTCOMES:
-Length of hospital stay. -Admission to ICU. - Blood transfusion (number of units of packes RBCs) -Angioembolization. -Surgery for uncontrolled recurrent bleeding. | 15 days

REFERENCES:
- [Background] Silverstein FE, Gilbert DA, Tedesco FJ, Buenger NK, Persing J. The national ASGE survey on upper gastrointestinal bleeding. I. Study design and baseline data. Gastrointest Endosc. 1981 May;27(2):73-9. doi: 10.1016/s0016-5107(81)73155-9. No abstract available. PMID 6971775
- [Background] Rockall TA, Logan RF, Devlin HB, Northfield TC. Incidence of and mortality from acute upper gastrointestinal haemorrhage in the United Kingdom. Steering Committee and members of the National Audit of Acute Upper Gastrointestinal Haemorrhage. BMJ. 1995 Jul 22;311(6999):222-6. doi: 10.1136/bmj.311.6999.222. PMID 7627034
- [Background] Elwakil R, Reda MA, Abdelhakam SM, Ghoraba DM, Ibrahim WA. Causes and outcome of upper gastrointestinal bleeding in Emergency Endoscopy Unit of Ain Shams University Hospital. J Egypt Soc Parasitol. 2011 Aug;41(2):455-67. PMID 21980783
- [Background] Quan S, Frolkis A, Milne K, Molodecky N, Yang H, Dixon E, Ball CG, Myers RP, Ghosh S, Hilsden R, van Zanten SV, Kaplan GG. Upper-gastrointestinal bleeding secondary to peptic ulcer disease: incidence and outcomes. World J Gastroenterol. 2014 Dec 14;20(46):17568-77. doi: 10.3748/wjg.v20.i46.17568. PMID 25516672
- [Background] Melcarne L, Garcia-Iglesias P, Calvet X. Management of NSAID-associated peptic ulcer disease. Expert Rev Gastroenterol Hepatol. 2016 Jun;10(6):723-33. doi: 10.1586/17474124.2016.1142872. Epub 2016 Mar 2. PMID 26775657
- [Background] Hwang JH, Fisher DA, Ben-Menachem T, Chandrasekhara V, Chathadi K, Decker GA, Early DS, Evans JA, Fanelli RD, Foley K, Fukami N, Jain R, Jue TL, Khan KM, Lightdale J, Malpas PM, Maple JT, Pasha S, Saltzman J, Sharaf R, Shergill AK, Dominitz JA, Cash BD; Standards of Practice Committee of the American Society for Gastrointestinal Endoscopy. The role of endoscopy in the management of acute non-variceal upper GI bleeding. Gastrointest Endosc. 2012 Jun;75(6):1132-8. doi: 10.1016/j.gie.2012.02.033. No abstract available. PMID 22624808
- [Background] Marmo R, Rotondano G, Piscopo R, Bianco MA, D'Angella R, Cipolletta L. Dual therapy versus monotherapy in the endoscopic treatment of high-risk bleeding ulcers: a meta-analysis of controlled trials. Am J Gastroenterol. 2007 Feb;102(2):279-89; quiz 469. doi: 10.1111/j.1572-0241.2006.01023.x. PMID 17311650
- [Background] Cheng HC, Sheu BS. Intravenous proton pump inhibitors for peptic ulcer bleeding: Clinical benefits and limits. World J Gastrointest Endosc. 2011 Mar 16;3(3):49-56. doi: 10.4253/wjge.v3.i3.49. PMID 21455342
- [Background] Sung JJ, Barkun A, Kuipers EJ, Mossner J, Jensen DM, Stuart R, Lau JY, Ahlbom H, Kilhamn J, Lind T; Peptic Ulcer Bleed Study Group. Intravenous esomeprazole for prevention of recurrent peptic ulcer bleeding: a randomized trial. Ann Intern Med. 2009 Apr 7;150(7):455-64. doi: 10.7326/0003-4819-150-7-200904070-00105. Epub 2009 Feb 16. PMID 19221370
- [Background] Sachs G, Shin JM, Howden CW. Review article: the clinical pharmacology of proton pump inhibitors. Aliment Pharmacol Ther. 2006 Jun;23 Suppl 2:2-8. doi: 10.1111/j.1365-2036.2006.02943.x. PMID 16700898
- [Background] Laine L, Shah A, Bemanian S. Intragastric pH with oral vs intravenous bolus plus infusion proton-pump inhibitor therapy in patients with bleeding ulcers. Gastroenterology. 2008 Jun;134(7):1836-41. doi: 10.1053/j.gastro.2008.03.006. Epub 2008 Mar 10. PMID 18423628
- [Background] Barkun AN, Herba K, Adam V, Kennedy W, Fallone CA, Bardou M. The cost-effectiveness of high-dose oral proton pump inhibition after endoscopy in the acute treatment of peptic ulcer bleeding. Aliment Pharmacol Ther. 2004 Jul 15;20(2):195-202. doi: 10.1111/j.1365-2036.2004.02035.x. PMID 15233700
- [Background] Sung JJ, Suen BY, Wu JC, Lau JY, Ching JY, Lee VW, Chiu PW, Tsoi KK, Chan FK. Effects of intravenous and oral esomeprazole in the prevention of recurrent bleeding from peptic ulcers after endoscopic therapy. Am J Gastroenterol. 2014 Jul;109(7):1005-10. doi: 10.1038/ajg.2014.105. Epub 2014 Apr 29. PMID 24777150